CLINICAL TRIAL: NCT02152787
Title: Comparison of Propofol 1mg/kg and Propofol 0.5mg/kg for Prevention of Emergence Agitation in Children Undergoing Strabismus Surgery During Sevoflurane Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3-2014-0028
Record Dates: First submitted 2014-05-28; First posted 2014-06-02 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Strabismus
Keywords: emergence agitation; propofol; strabismus surgery; children; elective strabismus surgery
MeSH Terms: conditions — Strabismus; Emergence Delirium | interventions — Propofol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1) propofol 1.0mg/kg group (Experimental): According to randomly allocated group, propofol 1.0mg/kg, propofol 0.5mg/kg or normal saline will be intravenously administered at the end of surgery
  Interventions: Drug: Injection of propofol 1.0mg/kg
- 2) propofol 0.5mg/kg group (Experimental): According to randomly allocated group, propofol 1.0mg/kg, propofol 0.5mg/kg or normal saline will be intravenously administered at the end of surgery
  Interventions: Drug: propofol 0.5mg/kg
- 3) normal saline group (Placebo Comparator): According to randomly allocated group, propofol 1.0mg/kg, propofol 0.5mg/kg or normal saline will be intravenously administered at the end of surgery
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Injection of propofol 1.0mg/kg
  Arms: 1) propofol 1.0mg/kg group
Drug: propofol 0.5mg/kg
  Arms: 2) propofol 0.5mg/kg group
Drug: normal saline
  Arms: 3) normal saline group

SUMMARY:
The occurrence of emergence agitation (EA) in pediatric patients who have received sevoflurane anesthesia is a common postoperative problem. Among various strategies for reducing the incidence and severity of EA, the use of pharmacological agents at the end of anesthesia is thought to be the most convenient and easily applicable method in clinical situation. The one of typical agents that can be administered in this way is propofol. Previous studies demonstrated that the use of propofol 1mg/kg at the end of anesthesia could reduce the incidence of EA with low incidence of postoperative nausea and vomiting. However, it was also demonstrated that the use of propofol 1mg/kg at the end of anesthesia could delay the emergence time. The purpose of this study is to compare the preventive effect on EA and the emergence time between propofol 1mg/kg and propofol 0.5mg/kg administered at the end of sevoflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. children (3-12 years old) scheduled for elective strabismus surgery undergoing general anesthesia.
2. ASA 1-2

Exclusion Criteria:

1. Patients with developmental disability, mental retardation, neurologic disorder, ongoing neurologic medication such as anticonvulsant, previously undergoing general anesthesia, a recent history of upper respiratory infection, parents difficult to read or understand the informed consent.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of the emergence agitation | from extubation up to 1 hour

SECONDARY OUTCOMES:
the emergence time | within the first 1hour after end of strabismus surgery
  The emergence time was defined as the time from discontinuation of sevoflurane to extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul, Seoul, South Korea